CLINICAL TRIAL: NCT03841643
Title: Comparison of Calcium Phosphate Cement With Patient-specific Implants for Cranial Reconstruction: a Randomized-controlled Trial
Brief Title: Comparison of Calcium Phosphate Cement With Patient-specific Implants for Cranial Reconstruction
Acronym: CRAN-PSI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Nathalie Neyt, maxillofacial surgeon, principal investigator, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2146
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Cranial Defect
Keywords: cranial reconstruction; cement; patient-specific implant; preprothetic surgery; atrophic jaw
MeSH Terms: interventions — Dental Bonding

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C group (Active Comparator): In the C group, the cranial bone defect will be reconstructed with HydrosetTM (Stryker, New Jersey, USA), calcium phosphate cement, according to the current standard practice at the department.
  Interventions: Device: cement
- P group (Experimental): In the P group, the cranial bone defect will be reconstructed with a patient-specific implant (KLS Martin, Tuttlingen, Germany).
  Interventions: Device: patient-specific implant

INTERVENTIONS:
Device: patient-specific implant — solid titanium implant that functions as a guiding template for harvesting, and as an implant for reconstruction of the cranial defect
  Arms: P group
Device: cement — norian cement for reconstruction of the cranial defect
  Arms: C group

SUMMARY:
Background Cranial reconstruction after monocortical bonegraft harvesting remains a clinical challenge for the maxillofacial surgeon. At present, there is no gold standard technique advised. Patient-specific implants are gaining terrain in the field of craniofacial reconstruction. Comparative studies on differences in success rates between different biomaterials for application in craniofacial surgery are lacking.

Aims The primary objective is to evaluate, in terms of cosmetic result, the postoperative successful outcome of patient-standardized implants for cranial reconstruction after bonegraft harvesting for jaw augmentation of patients with severely atrophic jaw.

Design Patients considered eligible for cranial bone-augmentation of the severely atrophic jaw, that provide their consent for participation in the trial, will be randomized at recruitment into either the patient-specific implant (P) or cement (C) group. In the P group, the cranial bone defect will be reconstructed with a patient-specific implant (KLS Martin, Tuttlingen, Germany). In the C group, the cranial bone defect will be reconstructed with HydrosetTM (Stryker, New Jersey, USA), calcium phosphate cement, according to the current standard practice at the department.

Parameters representing ease of application of the biomaterial , postoperative complication rate, cosmetic and functional outcome will be measured at fixed time-points during surgery and postoperative follow-up. A cone-beam computed tomography (CBCT) scan of both the donor (cranium) and receptor site (jaw) will be taken preoperatively, within 10 days postop, and 6 months post-operatively to measure biomaterial positioning.

Conclusions Systematic reviews demonstrate the need for randomized prospective studies regarding implantable biomaterials used in facial reconstructive surgery. We hypothesize that patient-specific implants provide more user-friendly alternatives to the standard care, with better cosmetic results.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older
* patients of all genders
* patients with moderate to extreme bone atrophy of the jaw, caused by periodontitis or edentulism
* patients requiring a full reconstruction (both anterior and posterior region)
* patients receiving their surgery and follow-up care at the AZ Sint-Jan Brugge-Oostende AV
* patients providing written informed consent

Exclusion Criteria:

* - Patients not eligible according to abovementioned criteria
* Patients with severe uncontrolled diabetes
* Patients with contraindications for general anesthesia
* Patients with known allergies to the biomaterials used
* Patients with cranial vault without diploe and/or cranial vault thickness <3mm, as defined with cone-beam CT
* Patients with previous surgery of the skull region
* Patients with an explicit risk of bleeding from cranial venous structures, as described by the radiologist based on his/her evaluation of the preoperative CBCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
volumetric measurement of cranial defect, through superimposition of the preoperative and postoperative cone beam computed tomography | within 10 days postoperative

SECONDARY OUTCOMES:
ease of application of both biomaterials, as graded with a 0 to 10 VAS score by the treating physician | perioperative
ease of application of both biomaterials, as determined by surgical time required | perioperative
postoperative complications, as graded by CTCAE 4.0 by the treating surgeon | within 30 days postoperative
patient satisfaction, as graded with a 0 to 10 VAS score | within 30 days postop
postoperative complications, as graded by CTCAE 4.0 by the treating surgeon | at 6 months postop
patient satisfaction, as graded with a 0 to 10 VAS score | at 6 months postop
final implant position, as determined with CBCT | at 6 months postop

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Neyt, MD, Principal Investigator — maxillofacial department, AZ Sint-Jan Brugge-Oostende AV
Locations (1):
- Department MKA, AZ Sint-Jan Brugge-Oostende AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No